CLINICAL TRIAL: NCT04753307
Title: Perioperative Inflammatory Response Assessment in High-risk Patients Undergoing Noncardiac Surgery - a Prospective Non-interventional Observational Study
Brief Title: Perioperative Inflammatory Response Assessment in High-risk Patients Undergoing Noncardiac Surgery
Acronym: INSIGHT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Christian Reiterer, PD Dr. med. univ., Medical University of Vienna
Other Study IDs: INSIGHT
Record Dates: First submitted 2021-02-03; First posted 2021-02-15 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Complications; Cardiovascular Complication; Myocardial Ischemia; Inflammation
MeSH Terms: conditions — Postoperative Complications; Myocardial Ischemia; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients at least 45 years at-risk for cardiovascular complications
  Interventions: Diagnostic Test: Laboratory measurements

INTERVENTIONS:
Diagnostic Test: Laboratory measurements — Inflammatory and cardiac biomarkers will be measured before surgery, and on the first, second, third and fifth postoperative day

SUMMARY:
Postoperative cardiovascular complications are common after noncardiac surgery. The association between perioperative inflammation and the occurrence of cardiovascular complications after surgery is still unknown. Therefore, we will evaluate as our primary aim the association between patients with increased postoperative inflammation, assessed with C-reactive protein measurements, and the occurrence of major cardiovascular complications after noncardiac surgery. We will further evaluate the influence of perioperative inflammation on the occurrence of postoperative acute kidney injury. We will also evaluate the association between inflammation and the influence on Days-At-Home within 30 days. Furthermore, we will evaluate the association between increased inflammatory biomarkers and postoperative N-terminal pro brain natriuretic peptide (NT-proBNP) concentration.

ELIGIBILITY:
All patients need to meet all of the following criteria for inclusion (1-4):

1. Surgery planned for more than two hours
2. ≥ 45 years of age
3. Provide written informed consent AND
4. Fulfill ≥ 1 of the following criteria (A-K)

Inclusion Criteria:

* NT-proBNP ≥ 200 ng/L
* Troponin T > 25 ng/L
* History of coronary artery disease
* History of peripheral artery disease (PAD)
* 75 years or older
* History of transient ischemic attack (TIA) or stroke
* Current smoking or cessation of smoking within 2 years
* Diabetes or currently taking anti-diabetic drug
* Hyperlipidemia
* History of hypertension or currently taking an antihypertensive drug
* Atrial fibrillation

Exclusion Criteria:

* Patients on immune-suppressive therapy
* ICU patients undergoing surgery
* Preoperative Sepsis/systemic inflammatory syndrome (SIRS) needing ICU treatment
* Preoperative hemodynamically instable patients, who require vasopressor or inotropic support
* History of severe heart failure (defined as left ventricular ejection fraction (LVEF) < 30%)
* Liver cirrhosis
* Chronic inflammatory bowel diseases (CIBD)
* Severe rheumatic diseases requiring immunosuppressive treatment

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at least 45 years and at-risk to develop postoperative cardiovascular complications undergoing noncardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiovascular complications | within 30 days after surgery and one year after surgery
  The primary aim of the study is to investigate the influence of the maximum C-reactive protein value (over the first 3 days after surgery) on the incidence of major cardiovascular complications within 30 days after surgery. The composite binary endpoint is defined as myocardial infarction, myocardial injury after noncardiac surgery, new onset of atrial fibrillation, stroke or death.

SECONDARY OUTCOMES:
C-reactive protein | within 30 days after surgery
  Secondary goals of the study are to investigate the influence of the C-reactive protein on day 5 on the incidence of cardiovascular complications within 30 days after surgery (combined binary endpoint).
Acute Kidney Injury - C-reactive proteint | within 5 days after surgery
  We will evaluate the influence C-reactive protein on the occurrence of postoperative acute kidney injury.
Acute Kidney Injury - Interleukin 6 | within 5 days after surgery
  We will evaluate the influence of Interleukin 6 on the occurrence of postoperative acute kidney injury.
Acute Kidney Injury - Procalcitonin | within 5 days after surgery
  We will evaluate the influence of Procalcitonin on the occurrence of postoperative acute kidney injury.
Acute Kidney Injury - Copeptin | within 5 days after surgery
  We will evaluate the influence of Copeptin on the occurrence of postoperative acute kidney injury.
Days at home within 30 days (DAH 30) | within 30 days after surgery
  We will evaluate the correlation between perioperative inflammation (C-reactive protein, Interleukin 6, Procalcitonin, Copeptin) and the number of days patient spend at home after surgery within 30 days (DAH30). Outcomes measure: Hospital discharge data will be used to calculate hospital length of stay. DAH30 will be calculated using mortality and hospitalization data from the date of the index surgery (day 0).
  For example, if a patient will die on day 2 after surgery, they were assigned 0 DAH30. If a patient will be discharged from hospital at day 6 after surgery but will be readmitted for 4 days before the second hospital discharge, we will assign 20 DAH30. If a patient will die within 30 days after surgery, irrespective of whether they will spend time at home, DAH30 will be scored as 0.
NT-proBNP | within 5 days after surgery
  We will evaluate the correlation of each of the following inflammatory parameters including C-reactive protein, Interleukin 6, Procalcitonin, Copeptin on postoperative NT-proBNP concentration. NT-proBNP will be measured before surgery, and on the first, second and third postoperative day.
Interleukin 6 | within 30 days after surgery
  We investigate the influence of the Interleukin 6 ,measured within the first five days after surgery, on the incidence of cardiovascular complications within 30 days after surgery (combined binary endpoint).
Copeptin | within 30 days after surgery
  We investigate the influence of the copeptin ,measured within the first five days after surgery, on the incidence of cardiovascular complications within 30 days after surgery (combined binary endpoint).
Procalcitonin | within 30 days after surgery
  We investigate the influence of the procalcitonin ,measured within the first five days after surgery, on the incidence of cardiovascular complications within 30 days after surgery (combined binary endpoint).

OTHER OUTCOMES:
Atrial fibrillation (AF) evaluation | within 5 days after surgery
  To evaluate the incidence of asymptomatic atrial fibrillation (AF) and symptomatic AF. Asymptomatic AF will be defined as irregular pulse without any clinical symptoms. Symptomatic AF will be defined as irregular pulse with one of the symptoms including racing heart, fluttering or palpitations; fatigue, shortness of breath; and lightheadedness.
SARS-Cov-2 - Inflammation | within first 5 days after surgery
  We will evaluate the effect of having a perioperative or previous infection with Severe Acute Respiratory Syndrome Corona Virus 2 (SARS-CoV-2) on postoperative inflammatory parameters including C-reactive protein, Copeptin, Interleukin 6 and Procalcitonin.
SARS-Cov-2 - Cardiovascular Complications | One year after surgery
  We will evaluate the effect of having a perioperative or previous infection with SARS-CoV-2 on the incidence of our composite outcome including myocardial myocardial infarction, myocardial njury after noncardiac surgery, new onset of atrial fibrillation, stroke or death.
  We will evaluate the outcome one year after surgery via a telephone interview.
SARS-Cov-2 One Year Follow-Up | One year after surgery
  We will evaluate the effect of a perioprative or previous SARS-Cov-2 infection on the neurocognitive function one year after surgery. Therefore, we will perform the telphone Montreal Cognitive Assessment (MoCA) before surgery and one year after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ridker PM, Luscher TF. Anti-inflammatory therapies for cardiovascular disease. Eur Heart J. 2014 Jul 14;35(27):1782-91. doi: 10.1093/eurheartj/ehu203. Epub 2014 May 26. PMID 24864079
- [Background] Kaptoge S, Seshasai SR, Gao P, Freitag DF, Butterworth AS, Borglykke A, Di Angelantonio E, Gudnason V, Rumley A, Lowe GD, Jorgensen T, Danesh J. Inflammatory cytokines and risk of coronary heart disease: new prospective study and updated meta-analysis. Eur Heart J. 2014 Mar;35(9):578-89. doi: 10.1093/eurheartj/eht367. Epub 2013 Sep 10. PMID 24026779
- [Background] Writing Committee for the VISION Study Investigators; Devereaux PJ, Biccard BM, Sigamani A, Xavier D, Chan MTV, Srinathan SK, Walsh M, Abraham V, Pearse R, Wang CY, Sessler DI, Kurz A, Szczeklik W, Berwanger O, Villar JC, Malaga G, Garg AX, Chow CK, Ackland G, Patel A, Borges FK, Belley-Cote EP, Duceppe E, Spence J, Tandon V, Williams C, Sapsford RJ, Polanczyk CA, Tiboni M, Alonso-Coello P, Faruqui A, Heels-Ansdell D, Lamy A, Whitlock R, LeManach Y, Roshanov PS, McGillion M, Kavsak P, McQueen MJ, Thabane L, Rodseth RN, Buse GAL, Bhandari M, Garutti I, Jacka MJ, Schunemann HJ, Cortes OL, Coriat P, Dvirnik N, Botto F, Pettit S, Jaffe AS, Guyatt GH. Association of Postoperative High-Sensitivity Troponin Levels With Myocardial Injury and 30-Day Mortality Among Patients Undergoing Noncardiac Surgery. JAMA. 2017 Apr 25;317(16):1642-1651. doi: 10.1001/jama.2017.4360. PMID 28444280
- [Background] Ridker PM, MacFadyen JG, Everett BM, Libby P, Thuren T, Glynn RJ; CANTOS Trial Group. Relationship of C-reactive protein reduction to cardiovascular event reduction following treatment with canakinumab: a secondary analysis from the CANTOS randomised controlled trial. Lancet. 2018 Jan 27;391(10118):319-328. doi: 10.1016/S0140-6736(17)32814-3. Epub 2017 Nov 13. PMID 29146124
- [Derived] Pichler A, Kurz A, Eichlseder M, Graf A, Eichinger M, Taschner A, Kabon B, Fleischmann E, Reiterer C; INSIGHT study group. PerIoperative iNflammatory reSponse assessment In hiGH-risk patienTs undergoing non-cardiac surgery (INSIGHT): study protocol of a prospective non-interventional observational study. BMJ Open. 2023 Jul 19;13(7):e065469. doi: 10.1136/bmjopen-2022-065469. PMID 37474184